CLINICAL TRIAL: NCT06436911
Title: Phase 1/2 Study to Evaluate Safety and Immunogenicity of a Prophylactic Plasmid DNA Booster Vaccine Against SARS-CoV-2 [Covigenix VAX-002] in Generally Healthy Adults 18 Years and Older
Brief Title: To Evaluate Safety and Immunogenicity of a Prophylactic Plasmid DNA
Acronym: VAX-002-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Entos Pharmaceuticals Inc. (Industry)
Collaborators: Calian CRO (Unknown); Q2 Solutions (Industry); PCI Pharma Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ENTVAX-002-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In Phase 1 up to 50 participants are planned to be randomized 1:1 into one of two groups: either 100 μg intramuscular (IM) injection or 250 μg IM injection. Participants are to receive a single 0.5 mL IM injection of VAX-002 100 μg or 250 μg on Day 0. Follow-up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180. An interim analysis is planned once all participants in Phase 1 have completed their Day 28 visit to evaluate dose-response and safety to support optimal dose selection for Phase 2.
  In Phase 2 approximately 250 participants will be enrolled and will receive a single 0.5 mL IM
  injection of the optimal VAX-002 dose (determined in the Phase 1 interim analysis) on Day 0. Follow- up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): In Phase 1 up to 50 participants are planned to be randomized 1:1 into one of two groups: either 100 μg intramuscular (IM) injection or 250 μg IM injection. Participants are to receive a single 0.5 mL IM injection of VAX-002 100 μg or 250 μg on Day 0. Follow-up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180. An interim analysis is planned once all participants in Phase 1 have completed their
  Interventions: Drug: COVIGENIX VAX- 002
- Phase 2 (Experimental): In Phase 2 approximately 250 participants will be enrolled and will receive a single 0.5 mL IM
  injection of the optimal VAX-002 dose (determined in the Phase 1 interim analysis) on Day 0. Follow- up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180.
  Interventions: Drug: COVIGENIX VAX- 002

INTERVENTIONS:
Drug: COVIGENIX VAX- 002 — ENTVAX-001-01

SUMMARY:
Currently, several vaccines are available to combat the COVID-19 pandemic. The persistence of SARS-CoV-2 globally requires the development of additional vaccines to aid in preventing further SARS-CoV-2 infections. Covigenix VAX-002 is a vaccine based off its predecessors VAX-001 and VAX-001-1b. All three are plasmid DNA vaccines that express key antigenic determinants from SARS-CoV-2 and use the Entos Pharmaceuticals' Fusogenix proteo-lipid vehicle (PLV) platform. Currently, the safety and tolerability of VAX-001 and VAX-001-1b for primary vaccination following 1 or 2 doses are being investigated in a Phase 1/2 study (ENTVAX01-101). In Phase 1, VAX-001 was administered to healthy adults on Day 0 and Day 14, as either 2 low doses (100 μg/dose) or 2 high doses (250 μg/dose). Overall, data suggest that VAX-001 is safe at both the low and high dose levels. The Phase 2 part evaluates VAX-001-1b in adults at a 100 μg dose level on a 1-dose and a 2-dose schedule (Days 0 and 28). An interim analysis conducted on data from 18 participants in the sentinel group who had received their first dose of 100 μg showed that VAX-001-1b was overall safe with minor adverse events (AEs) registered. No serious adverse events (SAEs) were reported. After a review of the data, the Data Safety Monitoring Committee (DSMC) provided their recommendations for the participants in the 100 μg dose sentinel group to receive a second dose.

The present study investigates the safety and immunogenicity of VAX-002 when given as a booster dose to generally healthy adults aged 18 years or older who have received a primary vaccination course or a booster dose of an authorized COVID-19 vaccine at least 3 months prior to Day 0.

VAX-002 was specifically designed to address the new circulating omicron variants of SARS-CoV-2.

The study consists of 2 parts: a dose-finding/safety evaluation part (Phase 1) to determine the dose of VAX-002 for booster vaccination (100 μg or 250 μg) followed by an adaptive Phase

DETAILED DESCRIPTION:
Phase 1 is the randomized, observer-blinded, multi-center, dose-finding part of the study, followed by an adaptive Phase 2 in which the optimal dose, determined from Phase 1, will be evaluated for safety and efficacy. In Phase 1 up to 50 participants are planned to be randomized 1:1 into one of two groups: either 100 μg intramuscular (IM) injection or 250 μg IM injection. Participants are to receive a single 0.5 mL IM injection of VAX-002 100 μg or 250 μg on Day 0. Follow-up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180. An interim analysis is planned once all participants in Phase 1 have completed their Day 28 visit to evaluate dose-response and safety to support optimal dose selection for Phase 2.

In Phase 2 approximately 250 participants will be enrolled and will receive a single 0.5 mL IM

injection of the optimal VAX-002 dose (determined in the Phase 1 interim analysis) on Day 0. Follow- up visits will occur on Days 7, 14, 17 (phone call visit), 21, 28, 42, and 180.

ELIGIBILITY:
Inclusion Criteria:

- 1. Generally healthy adults aged 18 years or older at the time of enrollment and with a body mass index (BMI) of ≤30 kg/m2

* Completion of a prior COVID-19 primary vaccination course or booster (any commercially available within the study country) at least 3 months prior to enrollment OR recent clinically documented SARS-CoV-2 infection (by polymerase chain reaction [PCR] or antibody test) in the past three months but not within one month from enrollment.
* Willing to refrain from receiving an authorized COVID-19 booster dose until at least 90 days post IP administration.
* Female participants of child-bearing potential must have practiced adequate contraception for 30 days before IP injection, have a negative pregnancy test on the day of IP injection, and agree to continue adequate contraception until 180 days after IP injection. (Please refer to Section 10.44 for the definition of childbearing potential and adequate contraception).
* Male participants must agree to continue adequate contraception until 180 days after IP injection.
* Able to consent to participate in the study and signed an Informed Consent Form (ICF).
* Able and willing to complete all the scheduled study procedures during the whole study period (approximately 6.5 months).
* Generally, in good health, as determined by a review of medical history and a physical examination within 14 days prior to IP injection.

Exclusion Criteria:

* 1. History of anaphylaxis to key ingredients within the vaccine. 2. History of seizure disorder, encephalopathy, or psychosis. 3. Female participant is pregnant (positive urine pregnancy test), lactating, or plans to become pregnant during the 180 days of enrollment. 4. Positive test result for human immunodeficiency virus (HIV) or hepatitis B and C at Screening (test to be performed at the discretion of the investigator based on medical history or physical examination). 5. Positive result of lateral flow test for SARS-COV-2 on Day 0. 6. Laboratory (hematological and biochemistry) examination that is out of normal range or greater than a Grade 2 abnormality. Grade 1 abnormalities will not be exclusionary if considered not clinically significant by the investigator. Laboratory tests include: complete blood count (CBC), prothrombin time (PT), partial thromboplastin time (PTT), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total bilirubin (T Bil), creatinine (CR), lipase, and blood glucose at screening. 7. Transient mild laboratory abnormalities may be rescreened once, and the participant will be excluded if the laboratory repeat test is abnormal as per local laboratory normal values and the investigator's assessment. 8. Presents with any acute febrile disease (oral temperature ≥37.5°C [99.5oF]) or active infectious disease within 48 hours prior to IP injection. 9. Unstable concomitant underlying conditions. Note: Stable condition defined as: the participant is appropriately managed on consistent disease management; for example, participants with well-controlled hypertension, adult-onset diabetes, benign prostate hypertrophy, or hypothyroid disease will be eligible for enrollment. The treatment regimen should be stable for at least 3 months prior to entering the study. Once IP treatment has started, the patient must be willing to maintain all aspects of the treatment regimen and forgo any elective changes in medication or management. Emergency changes in medication or management would be captured as an AE. 10. History of Guillain-Barre Syndrome or degenerative neurological disorders; a history of autoimmune, inflammatory disease or potential immune-mediated diseases (pIMD), or any condition that may put the participant at increased risk of safety events. 11. History of serious cardiovascular diseases, such as arrhythmia, conduction block, history of myocardial infarction, and severe hypertension not controlled with medication. 12. History of immunodeficiency, asplenia, or functional asplenia. 13. History of platelet disorder or other bleeding disorder that may cause contraindication for IM injection. 14. Heavy smoker (>10 cigarettes per day), vaper (>1 mL of e-liquid per day), or cannabis user ([near] daily use). Smokers have to agree to use the same cigarette brand throughout the study.

  15. History or diagnosis of coagulopathies. 16. Prior receipt of immunosuppressive medication, cytotoxic therapy, or systemic corticosteroids within 6 months before Day 0. 17. Recent receipt of blood products within 4 months before Day 0. 18. Administration of other investigational drugs within 3 months before Day 0 or planned use during the study period. 19. Currently has or a history of any condition that, in the opinion of the investigator, may interfere with the participant's compliance, evaluation of study objectives, or informed consent process (i.e., medical, psychological, social, or other conditions).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 13 months
  To evaluate the safety of VAX-002; Frequency and grade of each solicited local (injection site) and systemic reactogenicity AE from Day 0 through Day 28 Phase 2: Frequency and grade of each solicited local (injection site) and systemic reactogenicity AE at Day 0 through Day 28 Phase 1 only: Frequency and grade of unsolicited AEs, SAEs, and medically- attended AEs (MAAEs) from administration of investigational product (IP) through Day 28 Phase 2: Frequency and grade of unsolicited AEs, SAEs, and MAAEs from IP administration through Day 28 Phase 1/2: Frequency, type, and grade of SAEs related to IP administration, MAAEs related to IP administration, adverse events of special interest (AESI), or COVID-19 illness from IP administration through end-of-study (EOS)

SECONDARY OUTCOMES:
Secondary Outcome | 13 months
  To assess SARS-CoV-2 neutralizing antibody response:
  Phase 1 only : Antibody responses at specified timepoints from baseline (Day 0) through Day 28 - Geometric mean neutralizing antibody titers, as measured by SARS-CoV-2 neutralization assay
  Phase 1/2: Antibody responses at specified timepoints from baseline (Day 0) through EOS
  - Geometric mean neutralizing antibody titers, as measured by SARSCoV2 neutralization assay
  Phase 1 only: Seroconversion rate (% of participants who seroconvert), defined as a 4-fold or greater increase in neutralizing antibody titers, as measured by SARSCoV-2 neutralization assay from baseline (Day 0) through Day 28 Phase 1/2: Seroconversion rate (% of participants who seroconvert), defined as a 4-fold or greater increase in neutralizing antibody titers, as measured by SARS-CoV-2 neutralization assay at specified timepoints from baseline (Day 0) through EOS

OTHER OUTCOMES:
Exploratory Outcome | 13 months
  * To assess the humoral immune response Phase 1/2: Spot forming cells per million peripheral blood mononuclear cells (PBMC) and the differential expression of T cellular markers measured at specified timepoints from baseline (Day 0) through EOS Phase 1/2: Immunophenotyping flow cytometry performed at specified timepoints from baseline (Day 0) through EOS response of Covigenix VAX-002 booster to the SARS-CoV-2 S protein
  * To evaluate dose-response immunity
  * To evaluate antigen specific B and Tcell response by interferon-gamma enzyme-linked immunosorbent spot (ELISpot) assay with overlapping peptide pools (15mers overlapping by 11 residues) of vaccine antigens and by immunophenotyping T cells by flow cytometry (samples will be bio-banked for future analysis depending on the immune response)
  * To evaluate anti-fusion-associated small transmembrane (FAST) protein antibodies
  * To evaluate anti-dsDNA antibodies

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Centricity Research, Burlington, Ontario
  - Centricity Research, Toronto, Ontario
  - Diex Recherche Quebec, Québec, Quebec
  - Diex Recherche, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.entospharma.com/